CLINICAL TRIAL: NCT01169454
Title: Ventriculostomy in SAH: ICP Open or Not?
Brief Title: Ventriculostomy in Subarachnoid Hemorrhage (SAH): Intracranial Pressure (ICP) Open or Not?
Acronym: VISION 2
Status: Terminated | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00016054
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Cerebral Spinal Fluid; Ventriculostomy; Subarachnoid hemorrhage; Vasospasm; Human Subjects
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Monitor then drain: Subjects who are treated with intermittent CSF drainage
- Drain then monitor: Subjects who are treated with continuous CSF drainage at set pressure thresholds

SUMMARY:
The purpose of this study is to explore two currently accepted methods of intracranial pressure (ICP) management through cerebral spinal fluid (CRF) drainage for patients diagnosed with subarachnoid hemorrhage (SAH). This is a randomized observational study of two physician-prescribed approaches to managing ICP monitoring and CSF drainage for SAH patients. The study will enroll only those patients who have ICP monitoring. Because this is an observational study, there are no physical risks to the patient, the only risk is loss of confidentiality.

DETAILED DESCRIPTION:
Patients diagnosed with subarachnoid hemorrhage (SAH) who require intracranial pressure (ICP) management through cerebral spinal fluid (CRF) drainage will be eligible for this study.

Subjects will be randomized to receive one of two currently accepted methods of ICP management. The first is ICP monitoring with intermittent CSF drainage and the second is through continuous CSF drainage at set pressure thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Duke University NCCU
* Adult (18 years of age or older)
* Primary diagnosis is Subarachnoid Hemorrhage
* Intraventricular catheter in situ

Exclusion Criteria:

* Glasgow Coma Score = 3
* Hunt and Hess Score = 5
* Prisoners
* Ventriculostomy > 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cerebral artery vasospasm | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD RN CCRN, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Olson DM, Zomorodi M, Britz GW, Zomorodi AR, Amato A, Graffagnino C. Continuous cerebral spinal fluid drainage associated with complications in patients admitted with subarachnoid hemorrhage. J Neurosurg. 2013 Oct;119(4):974-80. doi: 10.3171/2013.6.JNS122403. Epub 2013 Aug 20. PMID 23957382